CLINICAL TRIAL: NCT02392442
Title: Pulmonary Effects of Bronchial Segmental Endotoxin Instillation in Humans
Brief Title: Effects of Bronchial Segmental Endotoxin Instillation in Humans
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 150091; 15-CC-0091
Record Dates: First submitted 2015-03-18; First posted 2015-03-19 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-05-16

CONDITIONS: Acute Lung Inflammation
Keywords: immunophenotypes; Bronchoalveolar Lavage; Bronchoscopy; Endotoxin Installation; niRNA
MeSH Terms: interventions — Sodium Chloride; Endotoxins

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 - Endotoxin (Experimental): 6 hour lavage post endotoxin
  Interventions: Biological: Endotoxin
- 2 - Endotoxin (Experimental): 24 hour lavage post endotoxin
  Interventions: Biological: Endotoxin
- 3 - Endotoxin (Experimental): 48 hour lavage post endotoxin
  Interventions: Biological: Endotoxin
- 4 Placebo comparator (Placebo Comparator): 6 hour control lavage
  Interventions: Other: Saline

INTERVENTIONS:
Other: Saline — Investigate the changes in miRNA signatures found in BAL and lung cells from healthy volunteers at baseline and at 6 hours after 1800 of normal Saline installed in six 30 mL aliquots into the left (lingual) and right (middle lobe) lung segments (360 mL total).
  Arms: 4 Placebo comparator
Biological: Endotoxin — Investigate the changes in miRNA signatures found in BAL and lung cells from healthy volunteers at baseline and at 6, 24, or 48 hours after endotoxin segmental lung challenge.
  Arms: 1 - Endotoxin; 2 - Endotoxin; 3 - Endotoxin

SUMMARY:
Background:

- When bacteria enter the lungs, serious infections can occur. Researchers want to learn more about the process of inflammation in the lungs by studying lung cells and the products that they make. Lung cells are influenced by infections, smoking, and molecules made within the body. Researchers also want to learn more about one of these molecules, called microRNA (or micro ribonucleic acid).

Objective:

- To better how the body responds to infection. Also, to understand which cells in the lung secrete microRNA and how they may influence other lung cells.

Eligibility:

- Healthy, non-smoking adults ages 18-45.

Design:

* Participants will be screened with a medical history and physical exam. They will have blood and urine tests and an electrocardiogram.
* Participants will have blood drawn from an arm vein. They will have an intravenous catheter (small plastic tube) placed in a vein.
* All participants will have bronchoscopy with bronchoalveolar lavage. They will be numbed with medicine. A thin flexible tube will be placed through the nasal passages or the mouth into the airways of the lung.

  * Some participants will have bronchoscopy with bronchoalveolar lavage (rinsing the airways with salt water) in order to obtain cells from lung. The water will then be suctioned out.
  * Some participants will have two bronchoscopies; during the first procedure, endotoxin, a molecule found in bacteria is squirted into a small portion of the lung. Endotoxin is a molecule that acts like an infection but isn t one. After 6 to 48 hours, bronchoscopy with with bronchoalveolar lavage will be done to look at the lung s response to endotoxin.
* Participants heart rhythm and rate, temperature and blood oxygen level will be monitored during the procedures.
* Participants will be called the next day to see how they are feeling.

DETAILED DESCRIPTION:
Defining the mechanisms that limit tissue injury during acute inflammation may provide the basis for preventing secondary organ dysfunction during serious infections. We plan to use the human endotoxin lung challenge model to study mechanisms associated with the initiation and resolution of lung inflammation.

Endotoxin (LPS), an outer membrane component of Gram-negative bacteria, is a major microbial factor that mediates inflammation associated with serious infections. For over fifty years, endotoxin has been administered to humans as a challenge agent in order to understand basic mechanisms of inflammation, to provide a proof of principle for pharmacologic interventions (e.g., anti-cytokines, corticosteroids), or as an adjuvant for immunotherapy of malignancies.

We previously developed a human model to study the initiation and resolution of inflammation in a lung segment following endotoxin bronchial instillation. The inflammatory response was limited to the challenged segment and had minimal associated systemic responses. After direct instillation into a lung segment, endotoxin elicits an inflammatory response characterized by the local production of inflammatory mediators, proteins and increases in cellularity. The predominate cell species found in the bronchoalveolar lavage (BAL) of the challenged segment changes from a neutrophil influx at 2 - 6 hours to an influx of monocytes and lymphocytes at 24 and 48 hours following endotoxin challenge. At 6 hours, BAL pro-inflammatory activity (i.e., tumor necrosis factor bioactivity and induction of intercellular adhesion molecule-1 on reporter cells) is present and absent at 24 and 48 hours post endotoxin. In addition, unique subsets of lymphocytes are present in the lung during this inflammatory response.

We have recently shown that non-cellular microRNAs (miRNAs) are present in archived BAL from normal healthy volunteer airways and are differentially expressed 6 hours after endotoxin-induced acute lung inflammation. miRNA are single stranded non-coding RNA that mediate posttranscriptional regulation of gene expression. Some extracellular miRNA species may modulate local and distant cell processes. miRNA can activate Toll-like receptors (TLRs) and have been described as blood biomarkers of different disease states. However, the specific role of extracellular or secreted miRNAs in the lung is poorly defined. Our research plan is designed to study the roles of miRNA in acute lung inflammation by investigating the changes in miRNA signatures found in BAL and lung cells from healthy volunteers at baseline and at 6, 24, or 48 hours after endotoxin segmental lung challenge. A panel of flow cytometry cell surface markers will be performed on blood and BAL cells and intracellular and secreted miRNA will be isolated from specific cell species (i.e., neutrophils, monocytes, macrophages, and lymphocytes). We hypothesize that miRNA will have a role in modulating the initiation and resolution of inflammation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Healthy 18 to 45 year old, nonsmoking subjects based on screening examination and laboratory tests.
  2. No significant active medical problems. This would include but not be limited to any cardiac disorder (e.g. arrhythmia, valvular heart disease), pulmonary disease (e.g. asthma requiring chronic medications, chronic bronchitis, emphysema), neurologic disorder (e.g.

     epilepsy), kidney disease (e.g. nephritis, nephrosis), rheumatologic disorder (e.g. inflammatory arthritis), endocrine disorder (e.g. diabetes, thyroid disease), liver disease (e.g. hepatitis), gastrointestinal disorder (e.g. inflammatory bowel disease) or infectious

     disease (e.g. human immunodeficiency virus).
  3. No concurrent medications including aspirin or non-steroidal anti-inflammatory drugs or have not taken these for at least 7 days prior to study participation.
  4. Previous smokers would have to have abstained from cigarettes for at least one year and have no greater than a 10-pack year smoking history. If you use a hookah, e-cigarette, or vaping more than once a week, you must abstain for at least 6 weeks prior to participating in the study.
  5. Females must be practicing active method of birth control or abstinence of sexual activity.
  6. Must be willing to have samples stored

EXCLUSION CRITERIA:

1. Any serious active medical problem as defined above
2. Pregnancy and/or lactation
3. BMI >30

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-06-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of cell-associated and secreted miRNA with specific types of resident and inflammatory cells in the lung. | 6, 24, or 48 hours after Endotoxin is instilled in the lung.
  Identification of cell-associated and secreted miRNA.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Suffredini, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent on IDP sharing.

REFERENCES:
- [Background] O'Grady NP, Preas HL, Pugin J, Fiuza C, Tropea M, Reda D, Banks SM, Suffredini AF. Local inflammatory responses following bronchial endotoxin instillation in humans. Am J Respir Crit Care Med. 2001 Jun;163(7):1591-8. doi: 10.1164/ajrccm.163.7.2009111. PMID 11401879
- [Background] Janssen O, Schaumann F, Holz O, Lavae-Mokhtari B, Welker L, Winkler C, Biller H, Krug N, Hohlfeld JM. Low-dose endotoxin inhalation in healthy volunteers--a challenge model for early clinical drug development. BMC Pulm Med. 2013 Mar 28;13:19. doi: 10.1186/1471-2466-13-19. PMID 23537365
- [Background] Sandstrom T, Bjermer L, Rylander R. Lipopolysaccharide (LPS) inhalation in healthy subjects increases neutrophils, lymphocytes and fibronectin levels in bronchoalveolar lavage fluid. Eur Respir J. 1992 Sep;5(8):992-6. PMID 1426208
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-CC-0091.html